CLINICAL TRIAL: NCT07074834
Title: Effectiveness of Metoprolol Succinate Combined With Trimetazidine in Reducing Inflammatory Biomarkers and Improving Clinical Outcomes in Coronary Heart Disease With Angina Pectoris
Brief Title: Metoprolol and Trimetazidine for Coronary Heart Disease With Angina
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shiyan City Renmin Hospital (Other Government)
Responsible Party: Principal Investigator, Qunxiong Fan, Principal investigator, Shiyan City Renmin Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: syrmyy2020-068
Record Dates: First submitted 2025-07-10; First posted 2025-07-20 (Actual); Last update posted 2025-07-20 (Actual); Status verified 2025-07

CONDITIONS: Coronary Heart Disease (CHD)
MeSH Terms: conditions — Coronary Disease | interventions — Trimetazidine

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental: Treatment Group (Experimental): Patients were randomized to receive routine drug therapy plus metoprolol succinate combined with trimetazidine for 3 months.
  Interventions: Drug: Metoprolol Succinate Sustained-Release Tablets; Drug: Trimetazidine; Drug: Routine Drug Therapy
- Active Comparator: Control Group (Active Comparator): Patients were randomized to receive routine drug therapy for 3 months.
  Interventions: Drug: Routine Drug Therapy

INTERVENTIONS:
Drug: Metoprolol Succinate Sustained-Release Tablets — Oral administration. Dose was 23.75 mg once daily for the first two weeks, then increased to 47.50 mg once daily.
  Arms: Experimental: Treatment Group
Drug: Trimetazidine — Oral administration. Dose was one tablet twice daily.
  Arms: Experimental: Treatment Group
Drug: Routine Drug Therapy — Included oral nitroglycerin tablets (0.5 mg twice daily), aspirin enteric-coated tablets (0.1 g once daily), and rosuvastatin calcium tablets (10 mg three times daily).

SUMMARY:
This is a prospective, randomized study to evaluate the effectiveness and safety of combining metoprolol succinate with trimetazidine compared to standard therapy for patients with coronary heart disease (CHD) and angina pectoris. The study aims to assess the effects of the combination therapy on inflammatory biomarkers, clinical efficacy, angina symptoms, and left ventricular function over a 3-month treatment-period.

DETAILED DESCRIPTION:
Coronary heart disease (CHD) with angina pectoris is a significant cause of morbidity and mortality. While standard treatments like β-blockers (e.g., metoprolol succinate) are effective, many patients continue to experience symptoms. Inflammation is known to play a crucial role in the pathophysiology of CHD. This study was designed to investigate whether the addition of trimetazidine, a myocardial anti-ischemic agent that improves cellular energy metabolism, to standard metoprolol succinate therapy could offer superior benefits. This prospective study enrolled and randomized 102 patients with CHD and angina into two groups: a control group receiving routine drug therapy and a treatment group receiving routine therapy plus metoprolol succinate and trimetazidine. The primary objective was to compare the therapeutic efficacy, changes in angina attack frequency and severity, improvements in left ventricular function, and reductions in key inflammatory markers (IL-1β, TNF-α, hs-CRP, IL-18) between the two groups after 3 months of treatment. The study aims to provide evidence for this combination therapy as a safe and effective option for managing CHD with angina pectoris.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of CHD and angina pectoris based on CAD and angina pectoris guidelines.
* History of previous myocardial infarction, confirmed by coronary angiography or coronary computed tomography angiography, with at least one coronary artery stenosis ≥50%.
* Disease duration over 3 months.
* Frequency of angina attacks in the past week was ≥3 times, with a severity grade of I, II, or III.
* All patients signed an informed consent form.

Exclusion Criteria:

* Patients with mental disorders, drug allergies, acute myocardial infarction, electrolyte imbalances, important organ dysfunction, or cardiomyopathy.
* Patients with severe immune or infectious diseases.
* Those with stable symptoms or no symptoms after acute coronary syndrome.
* Patients with severe arrhythmia, uncontrolled hypertension (SBP ≥180 mmHg or DBP ≥110 mmHg), pacemaker, or aortic dissection.
* Pregnant or lactating women.
* Patients requiring revascularization (e.g., multi-vessel disease, left main disease, or ischemic areas >10% of the left ventricle).
* Patients who participated in other clinical trials within the past month.

Ages: 46 Years to 76 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2021-02-01 (Actual); Primary Completion 2022-09-30 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Change in Clinical Efficacy Rate | At 3 months
  Clinical efficacy was assessed based on symptom changes and reduction in angina attacks. Efficacy was categorized as "Marked effect" (symptoms nearly controlled, attacks decreased >80%), "Effective" (symptoms partially improved, attacks decreased 50-80%), or "Ineffective". The total effective rate was calculated as (Marked effect + Effective) / Total cases × 100%.
Change in Frequency of Angina Attacks | From Baseline to 3 months
  The mean number of angina attacks per week was recorded and compared between groups.
Change in Serum Inflammatory Markers | From Baseline to 3 months
  Changes in serum levels of Interleukin-1 beta (IL-1β), Tumor Necrosis Factor-alpha (TNF-α), and high-sensitivity C-reactive protein (hs-CRP) were measured using ELISA and immune transmission nephelometry.

SECONDARY OUTCOMES:
Change in Angina Pain Score | From Baseline to 3 months
  Pain severity was assessed using the Visual Analog Scale (VAS) with a score from 0 (no pain) to 10 (most severe pain).
Change in Duration of Angina Episodes | From Baseline to 3 months
  The mean duration of angina attacks was recorded and compared.
Change in Left Ventricular Ejection Fraction (LVEF) | From Baseline to 3 months
  LVEF was measured by color Doppler ultrasound to assess left ventricular systolic function.
Change in Left Ventricular End-Diastolic Diameter (LVEDD) | From Baseline to 3 months
  LVEDD was measured by color Doppler ultrasound to assess cardiac remodeling.
Change in Left Ventricular End-Systolic Diameter (LVESD) | From Baseline to 3 months
  LVESD was measured by color Doppler ultrasound to assess cardiac remodeling.
Change in Serum Interleukin-18 (IL-18) levels | From Baseline to 3 months
  Serum IL-18 levels were measured using ELISA.
Incidence of Adverse Reactions | Over 3 months
  The number and percentage of patients experiencing adverse reactions, including gastrointestinal abnormalities, arrhythmias, or hypotension, were recorded.

CONTACTS AND LOCATIONS:
Locations (1):
- Renmin Hospital, Hubei University of Medicine, Shiyan, Hubei, China